CLINICAL TRIAL: NCT07363694
Title: AN INTERVENTIONAL PHASE 2/3, RANDOMIZED, DOUBLE-BLIND, THIRD PARTY-UNBLINDED, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY TO INVESTIGATE EFFICACY AND SAFETY OF PF-07275315 IN ADULT PARTICIPANTS WITH MODERATE-TO-SEVERE CHRONIC OBSTRUCTIVE PULMONARY DISEASE (COPD)
Brief Title: A Study to Learn About the Study Medicine Called PF-07275315 in People With Moderate to Severe Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4531031; 2024-518587-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2026-01-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All dosing syringes will be masked and an unblinded administrator will administer the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 2 Treatment Arm A (Experimental)
  Interventions: Drug: PF-07275315 dose 1
- Phase 2 Treatment Arm B (Experimental)
  Interventions: Drug: PF-07275315-dose 2
- Phase 2 Treatment Arm C (Placebo Comparator)
  Interventions: Drug: Placebo
- Phase 3 Treatment Arm A (Experimental)
  Interventions: Drug: PF-07275315-dose 3
- Phase 3 Treatment Arm B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07275315 dose 1 — SC injection dose 1
  Arms: Phase 2 Treatment Arm A
Drug: PF-07275315-dose 2 — SC injection dose 2
  Arms: Phase 2 Treatment Arm B
Drug: Placebo — SC injection matched
  Arms: Phase 2 Treatment Arm C; Phase 3 Treatment Arm B
Drug: PF-07275315-dose 3 — SC injection dose 3
  Arms: Phase 3 Treatment Arm A

SUMMARY:
The purpose of this clinical trial is to learn about the effects and safety of the study medicine PF-07275315 for the potential treatment of COPD. COPD is a condition that makes it difficult to breathe, which negatively impacts the quality of life and functioning of people who are affected.

This study is seeking participants who:

* Are 35 to 80 years old
* Have had moderate-to-severe COPD for at least 12 months
* Have a documented history of at least 2 moderate or severe exacerbations within the last 12 months
* Have been continuously taking their regular maintenance treatment(s) for COPD over at least 6 months at a stable dose for 3 months

All participants will receive PF-07275315 or a placebo. A placebo does not have any medicine in it but looks just like the medicine being studied.

PF-07275315 or placebo will be given as multiple shots in the clinic over the course of 24 weeks for the Phase 2 part and 52 weeks for the Phase 3 part. We will compare the results of people receiving PF-07275315 to those of the people who do not. This will help us determine if PF-07275315 is safe and effective.

Participants who will be involved in the Phase 2 part of the study for about 40 weeks. During this time, they will have 11 visits at the study clinic.

Participants who will be involved in the Phase 3 part of the study for about 68 weeks. During this time, they will have 18 visits at the study clinic.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) for at least 12 months (based on Global Initiative for Chronic Obstructive Lung Disease [GOLD] definition).
* Spirometry values (post-bronchodilator forced expiratory volume in 1 second [FEV1]/forced vital capacity [FVC] less than [<] 70 percent (%) and post-bronchodilator FEV1 % predicted <70%, but greater than equal to 30%).
* Continuous treatment with standard of care triple therapy of LABA + LAMA + ICS for ≥ 6 months prior to Screening Visit 1 and at a stable dose for ≥3 months
* Documented history of at least 2 moderate or severe ECOPD within the last 12 months prior to Screening.

Key Exclusion Criteria:

* Significant pulmonary disease other than COPD.
* Requirement for continuous chronic treatment with oxygen at >4.0 liters / minute by nasal cannula or equivalent.
* Hypoxemia with a resting SpO2 <88% while breathing ambient air (or on the participant's usual level of oxygen supplementation).
* Clinically significant cardiovascular disease, acute and/or severe left heart failure, or heart failure partial ejection fraction, and/or cor pulmonale.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1156 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2030-10-24 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
Phase 2 part: Change from baseline in pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 24 | Baseline to Week 24
  FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV1 is obtained from spirometry.
Phase 3 part: Annualized rate of moderate or severe ECOPD | Baseline to Week 52
  Exacerbation of Chronic Obstructive Pulmonary Disease (ECOPD) are sudden worsening of respiratory symptoms that significantly worsen lung function and quality of life.

SECONDARY OUTCOMES:
Phase 2: Annualized rate of moderate or severe ECOPD. | Baseline to Week 24
Phase 2: Change from baseline in pre-BD FEV1 up to Week 24. | Baseline to Week 24
Phase 2: Change from baseline in trough, pre- and post-BD FEV1 up to Week 24 | Baseline to Week 24
Phase 2: Change from baseline in trough, pre- and post-BD FVC and FEV1/FVC ratio, % predicted FEV1, % predicted FVC up to Week 24. | Baseline to Week 24
Phase 2: Change from baseline in trough FEV1 responsiveness to BD up to Week 24. | Baseline to Week 24
Phase 2: Incidence and severity of TEAEs throughout Phase 2 part of the study. | Baseline to Week 24
Phase 2: Incidence of treatment-emergent adverse events and serious adverse events leading to discontinuation. | Baseline to Week 24
Phase 2: Incidence of clinical abnormalities in clinical laboratory values, ECG measurements, and vital signs. | Baseline to Week 24
Phase 3: change from baseline in pre- and post-BD FEV1 at Week 12 and Week 52. | Baseline to Week 52
Phase 3: Percentage of participants with ≥4 points improvement from baseline in Saint George's Respiratory Questionnaire (SGRQ) score at Week 52. | Baseline to Week 52
Phase 3: Percentage of participants with ≥2 points improvement from baseline in the COPD Assessment Test (CAT) total score at Week 52. | Baseline to Week 52
Phase 3: Percentage of participants with ≥2 points improvement from baseline in E-RS:COPD total score at Week 52. | Baseline to Week 52
Phase 3: Annualized rate of severe ECOPD. | Baseline to Week 52
Phase 2: Change from baseline of clinical abnormalities in clinical laboratory values, ECG measurements, and vital signs. | Baseline to Week 24
Phase 3: Annualized rate of exacerbations requiring emergency department visit and/or hospitalization. | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - NewportNativeMD, Inc., Newport Beach, California
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Reed Medical Research, Miami, Florida
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - Salem Chest Specialists, Winston-Salem, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Clinical Research Associates of Central PA, LLC, DuBois, Pennsylvania
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Premier Research Center, LLC, Hendersonville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4531031